CLINICAL TRIAL: NCT00997620
Title: A Double Blind, Placebo Controlled Randomized Trial Evaluating the Effects of Fluticasone Nasal Spray in Subjects With Seasonal Allergic Rhinitis and a History of Sleep Disturbance on Cognitive Performance and Daytime Sleepiness
Brief Title: Fluticasone Furoate Treatment of Daytime Somnolence and Cognitive Performance in Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Western Sky Medical Research (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Lyndon Mansfield, Director, Western Sky Medical Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2008-4
Record Dates: First submitted 2009-10-15; First posted 2009-10-19 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Hay Fever; Daytime somnolence; Cognition
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Disorders of Excessive Somnolence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo treatment given as a once daily dose intranasally.in subjects with active seasonal allergic rhinitis.
  Interventions: Drug: Placebo
- Fluticasone Furoate (Experimental): IFluticasone Furoate 110 mcg given intranasly once daily in am as an active treatment of seasonal allergic rhinitis
  Interventions: Drug: Fluticasone furoate Nasal Spray 110 mcg

INTERVENTIONS:
Drug: Fluticasone furoate Nasal Spray 110 mcg — Fluticasone fuorate nasal spray 110 mcg 2 sprays each nostril am will be compared to similar appearing placebo given 2 sprays each nostril am. The subjects will receive one week placebo nasal spray to establish a baseline then they will then be switched to a nasal spray of fluticasone furoate 110 mcg once daily and continue the evaluations.
  Other Names: Fluticasone Furoate Nasal Spray
  Arms: Fluticasone Furoate
Drug: Placebo — Fluticasone nasal spray 2 sprays each nostril will be compared to similar appearing placebo. The subjects will receive one week placebo nasal spray to establish a baseline then they will then be switched to a nasal spray of Placebo once daily and continue the evaluations.
  Other Names: Placebo Veramyst Nasal Spray
  Arms: Placebo

SUMMARY:
The hypothesis is that treating hay fever patients who had daytime sleepiness and slowed thinking because of the hay fever will improve when treated with an effective anti-hay fever medication, an intranasal steroid, that is will have less daytime sleepiness and demonstrate better thinking.

DETAILED DESCRIPTION:
In this study of patients with seasonal allergic rhinitis we will monitor daytime sleepiness as measured by validated daytime sleep score (Eppworth Daytime Sleepiness Scale) and cognitive performance weekly as measured by a validated test of cognitive performance (TOVA). The treatment group with intervention of fluticasone furoate nasal spray 110 mcg two sprays in each nostril once daily will be compared to a placebo treated group of similar subjects with seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic seasonal allergic rhinitis symptoms for at least 2 years at the time of study in the season of the study.
* Allergy skin tests positive for the airborne allergens present at the study time within the past 12 months.
* A score of 2 or more on the NRQLQ of the Rhinitis Quality of LIfe Questionnaire.
* Active allergic rhinitis on 4 of 7 days during run-in week, and evidence on sleep scales of drowsiness on 3 of 7 days.
* Ability to read, understand and give informed consent.
* Ability to understand and carry out responsibilities of the study

Exclusion Criteria:

* Any chronic disease or other acute disease, which could influence central nervous system.
* The use of any medication, which could affect central nervous system function.
* Unwillingness to participate in the study.
* Inability to understand testing procedures or use of medication.
* Hypersensitivity to fluticasone or vehicle of nasal sprays.
* Any sleep disorders including obstructive sleep apnea.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided
This a single study site and at end IPD will be used in analyis by PI

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo for comparison
  Placebo: Fluticasone nasal spray 2 sprays each nostril will be compared to similar appearing placebo
- Fluticasone Furoate: Active treatment
  Fluticasone furoate Nasal Spray: Fluticasone nasal spray 2 sprays each nostril will be compared to similar appearing placebo
Period: Overall Study
Arm/Group | Placebo | Fluticasone Furoate
Started | 19 | 21
Completed | 19 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fluticasone Furoate | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Full Range); unit: years] | 36 [18 to 55] | 38 [19 to 55] | 37 [18 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Performance on Test of Variables of Attention (TOVA) - a Standardized Test of Cognitive Performance
Description: The outcomes measures for TOVA are errors of omission. Targets which were not identified. Errors of commission are when targets are identified incorrectly. Reaction time is reported as the average time in milliseconds for the responses. The results are reported as mean and standard deviation as baseline and after 2 weeks of intervention. The difference between the means was evaluated by paired t testing.
Time Frame: over 2 weeks
Measure: Mean (Standard Deviation); unit: number of errors
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 19 | 21
number of errors
  Baseline | 2.63 (2.98) | 3.95 (3.18)
  After 2 weeks intervention | 1.20 (1.24) | 1.83 (1.90)

2. Primary Outcome: Performance on Test of Variables of Attention (TOVA) - a Standardized Test of Cognitive Performance, Errors of Commission.
Description: The outcomes measures for TOVA are errors of commission. Targets which were identified incorrectly. Targets which are not identified, errors of omission and average time of each target viewing.
Time Frame: after 2 weeks intervention
Measure: Mean (Standard Deviation); unit: non identified targets
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 19 | 21
non identified targets
  Baseline | 2.33 (4.54) | 1.54 (3.72)
  After 2 weeks intervention | 5.75 (14.10) | 1.58 (4.11)

3. Primary Outcome: Performance on Test of Variables of Attention (TOVA) - a Standardized Test of Cognitive Performance, Response Time for Targets.
Description: The outcomes measures for TOVA are the length of time to respond to targets. The time function represents the average time spent in milliseconds spent on each target.
Time Frame: over 2 weeks
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 19 | 21
milliseconds
  Baseline | 387.58 (77.03) | 363.38 (61.91)
  After 2 weeks intervention | 412.47 (66.16) | 391.81 (91.41)

4. Secondary Outcome: Change in Epworth Sleep Scale
Description: The Epworth sleepiness scale measures is a validated test of daytime sleepiness which involved the subjects answering 8 questions. Each question is answered on a 0 - 3 scale with 3 being the most likely associated with drowsiness. The score is reported as a composite score of 8 questions, with a minimum score of 0 and a maximum score of 24. A higher composite score represents more likelihood of daytime sleepiness. It is administered between 1500 and 1700 daily.
Time Frame: Baseline and after 2 weeks intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 19 | 21
units on a scale
  Baseline | 13.28 (3.42) | 13.83 (3.82)
  After 2 weeks intervention | 12.80 (4.10) | 10.80 (5.48)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; The statistical analysis was of t testing of the difference of the mean between the baseline and after two weeks. The power analysis was prior to data collection was not performed for this test. The null hypothesis is no different, no difference between placebo and active treatment; Test type: Other; p < .05, t-test, 2 sided; Mean Difference (Net) = 0.50

5. Secondary Outcome: Change From Baseline in Nocturnal Rhinoconjunctivitis Quality of Life Questionaire
Description: In nocturnal rhinoconjunctivitis quality of life questionnaire instrument to measure the effects of nasal disorder on nighttime sleep and awakening. It consists of 16 questions. The scale is from 0-6, 0 being not troubled and 6 reflecting extreme trouble. This survey is interpreted as a minimal clinically important difference of each question. A change of +/- 0.5 is a threshold of minimally important clinical difference. Higher value mean more disturbance.
Time Frame: 2 weeks
Population: The NRQLQ values represent the average for each intervention.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo Nasal Spray: One week placebo nasal spray followed by two weeks placebo nasal spray.
- Fluticasone Furoate Nasal Spray: One week placebo nasal spray followed by two weeks fluticasone furoate nasal spray.
Arm/Group | Placebo Nasal Spray | Fluticasone Furoate Nasal Spray
Number analyzed (Participants) | 19 | 21
units on a scale
  Difficulty getting to sleep | -0.158 (.384) | -0.67 (0.326)
  Unable to get a good nights sleep | -0.579 (0.369) | -0.904 (0.389)
  Restless (tossing and turning) | -0.789 (0.329) | -0.90 (0.37)
  Having to get up because of stuffy nose. | -0.632 (0.298) | 1.49 (3.01)
  Nasal congestion | -0.7894 (0.329) | -0.76 (0.44)
  Sinus pressure or pain | -0.738 (0.389) | 1.569 (4.2494)
  Runny nose | -0.895 (0.252) | -0.429 (0.405)
  Post-nasal drip | -1.2105 (0.493) | -1.333 (0.380)
  Headache | -1.105 (0.431) | -1.3 (0.576)
  Feel tired and unrefreshed | -1.158 (0.448) | -0.286 (0.962)
  Nasal congestion or stuffy nose | -0.684 (0.380) | -0.857 (0.340)
  Congestion in sinuses | 0.05 (0.354) | -1.048 (0.297)
  time to clear nighttime drainage after waking | -0.474 (0.299) | -1.190 (0.418)
  Need to rub nose or eyes | -0.053 (0.0291) | -1.4286 (0.369)
  Have to take medication | -0.474 (0.337) | -1.429 (0.434)
  Having to avoid symptom triggers | -0.474 (0.345) | -1.190 (0.541)

6. Secondary Outcome: Nasal Symptom Scores
Description: Total nasal symptom score was measured AM and PM. The reflective scale measures subjective symptoms over the previous 12 hours. Instantaneous symptoms measure how subjects felt at the present time. The score consists of subjective perception of nasal congestion, rhinorrhea, nasal itching and sneezing. The scale for each symptom is 0 - not present, 1- mild (present but minimal), 2 - moderate (symptoms are bothersome but tolerable), 3 - severe (symptoms are not tolerable). The baseline value was the mean of the 7 day placebo run-in for the combined scores. This was calculated for the placebo group and the fluticasone group for both the instantaneous and the reflective scores. The intervention time utilized the same combined AM and PM reflective and instantaneous scoring. The data was analyzed using two sample t test comparison of the placebo vs fluticasone furoate group. Low value, less symptoms. High value, more symptoms. Minimum score is 0. Maximum score is 24.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Nasal Spray | Fluticasone Furoate Nasal Spray
Number analyzed (Participants) | 19 | 21
units on a scale
  Instaneous Baseline | 12.65 (4.9) | 12.88 (4.26)
  Instaneous Post 2 Weeks Therapy | 13.74 (4.52) | 10.84 (6.34)
  Reflective Baseline | 13.53 (4.4) | 12.99 (3.73)
  Reflective Post 2 Weeks Therapy | 14.02 (4.65) | 11.19 (6.05)

ADVERSE EVENTS:
Arm/Group | Placebo | Fluticasone Furoate
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No